CLINICAL TRIAL: NCT05245292
Title: An Open Label, Single Arm Study of the Safety and Antiretroviral Activity of Two Long-acting Broadly Neutralizing Antibodies Plus an IL-15 Superagonist in ART-treated Adults Living With HIV During Analytical Treatment Interruption
Brief Title: 3BNC117-LS and 10-1074-LS Plus N-803 (bNAb+N-803)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Weill Medical College of Cornell University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCA-1031 (ES38918); 1U01AI145921 (NIH)
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: 3BNC117-LS; 10-1074-LS; Broadly Neutralizing Antibody; N-803; IL-15 superagonist complex
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Broadly Neutralizing Antibodies; Antibodies, Monoclonal; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3BNC117-LS + 10-1074-LS + N-803 (Experimental): 3BNC117-LS dosed at 30 mg/kg IV, day 0 10-1074-LS dosed at 10 mg/kg IV, day 0 N-803 dosed at 6 mcg/kg, SC, 8 doses every 3 weeks (week 1 through week 22)
  Interventions: Drug: 3BNC117-LS; Drug: 10-1074-LS; Drug: N803

INTERVENTIONS:
Drug: 3BNC117-LS — Intravenous infusion of 3BNC117-LS at 30 mg/kg
  Other Names: broadly neutralizing antibody; monoclonal antibody
Drug: 10-1074-LS — Intravenous infusion of 10-1074-LS at 10 mg/kg
  Other Names: broadly neutralizing antibody; monoclonal antibody
Drug: N803 — Subcutaneous injections of N803 at 6 mcg/kg
  Other Names: IL-15 superagonist complex

SUMMARY:
The proposed study is a phase 1, open label, single arm study to evaluate the safety and antiretroviral activity of the combination of two long-acting broadly neutralizing antibodies, 3BNC117-LS dosed once at 30 mg/kg and 10-1074-LS dosed once at 10 mg/kg, both intravenously (IV) at week 0, plus an IL-15 superagonist complex, N-803, dosed at 6 mcg/kg, subcutaneously (SC) at week 1 and then every 3 weeks for a total of 8 doses, in ART-treated adults living with HIV during analytical treatment interruption.

DETAILED DESCRIPTION:
The proposed study is a phase 1, open label study of the safety and antiretroviral activity of the 3BNC117-LS plus 10-1074-LS broadly neutralizing antibody (bNAb) combination plus N-803, an IL-15 superagonist complex, in ART-treated individuals living with HIV during interruption of ART.

Thirty-six eligible participants will be enrolled sequentially and will be assigned to Group A or Group B after Monogram PhenoSense Assay results become available: Group A - participants with 3BNC117 and 10-1074 IC90 less or equal to 1 mcg/mL and MPI greater or equal to 98% by the Monogram PhenoSense assay using PBMCs; Group B - all other participants, including participants from whom the PhenoSense Assay (PBMC) does not yield a result.

Participants will discontinue ART on day 2 (2 days after the first antibody infusions) and will be followed for up to 72 weeks while off ART and for 12 weeks after ART is resumed.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, age 18 to 70.
2. Confirmed HIV-1 infection.
3. On antiretroviral therapy with plasma HIV-1 RNA levels of < 50 copies/ml and no reported interruption of ART for 7 consecutive days or longer for at least 48 weeks, and < 20 copies/ml at screening.

   NOTE: At least two Viral Load (VL) measurements within 48 weeks prior to the Step 0 screening visit must be available for review. A single plasma HIV-1 RNA > 50 copies/mL but < 200 copies/mL that is followed by an HIV-1 RNA <50 copies/mL is permitted.
4. Current CD4+ T cell counts > 450 cells/mcL, CD4+ T cell % ≥ 15%, and CD4+ T cell count nadir of ≥ 200 cells/mcL.
5. If on an NNRTI-based regimen, willing to switch to an integrase inhibitor-based regimen for at least 4 weeks prior to discontinuing ART.
6. For participants who can become pregnant (i.e., participants who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy), negative pregnancy test at screening (Step 0) and within 48 hours prior to day 0 (Step 1 entry).
7. Participants who can become pregnant must agree to use two methods of contraception, one of which must be from the highly effective methods for contraception listed below. Barrier methods of contraception are permitted for the second method of contraception. Contraception must be used from 10 days prior to the first of the investigational products (IP), while receiving the IPs, for 12 months after the last IP dose and until ART is reinitiated and viral suppression is achieved.
8. Participants who can impregnate a partner and who are engaging in sexual activity that could lead to pregnancy must agree to use condoms from 10 days prior to the first dose of the investigational products (IP), while receiving the IPs, and for 12 months after the last IP dose to avoid impregnating a partner who can get pregnant.
9. Willingness to use barrier protection (male or female) during sexual activity during analytical treatment interruption (ATI) and until viral re-suppression for those who re-start ART.

Exclusion Criteria:

1. History of AIDS-defining illness within 3 years prior to enrollment.
2. History of systemic corticosteroids (e.g. an equivalent dose of prednisone of > 20 mg daily for > 14 days), immunosuppressive anti-cancer, interleukins, systemic interferons, systemic chemotherapy or other medications considered significant by the trial physician within the last 6 months.
3. Any clinically significant acute or chronic medical condition (e.g. such as autoimmune diseases, cirrhosis), other than HIV infection, that in the opinion of the investigator would preclude participation.
4. History of or current clinical atherosclerotic cardiovascular disease (ASCVD), as defined by 2013 ACC/AHA guidelines.
5. QTcF interval ≥ 440 ms at screening.
6. Any history of an HIV-associated malignancy, including Kaposi's sarcoma, or any type of lymphoma or virus-associated cancers.
7. History of Progressive Multifocal Leukoencephalopathy (PML).
8. Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months;
9. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood.
10. Participants with known hypersensitivity to any constituent of the investigational products.
11. Pregnancy or lactation.
12. ART initiated during acute infection (defined as p24, HIV NAAT, or HIV RNA PCR positive, and negative or indeterminate HIV antibody testing).
13. Receipt of cabotegravir-LA IM or rilpivirine-LA IM within 24 months prior to Step 1 study entry.
14. Known resistance to all drugs within two or more ARV drug classes.
15. Laboratory abnormalities in the parameters listed below:

    * Absolute neutrophil count < 1,000 cells/microlitre;
    * Hemoglobin < 10 gm/dL;
    * Platelet count < 100,000 cells/microlitre;
    * ALT > 1.5 x ULN;
    * AST > 1.5 x ULN;
    * Total bilirubin > 1.5 x ULN;
    * eGFR < 60 mL/min/1.73m2;
16. Any history of receipt of therapeutic HIV vaccine or HIV monoclonal antibody therapy.
17. Participation in any clinical study of an investigational product within 12 weeks prior to study entry (day 0) or expected participation in such a study during this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related Grade 3 adverse events and serious adverse events | 72 weeks
  The number of participants with treatment-related solicited and unsolicited grade 3 and serious adverse events (including confirmed laboratory abnormalities), or premature study treatment discontinuation due to an adverse event (regardless of grade).
Any serious adverse events | 72 weeks
  The number of participants with serious adverse events, regardless of relationship to 3BNC117-LS, 10-1074-LS and N-803.
Dosing completion | 24 weeks
  The proportion of participants who complete dosing with 3BNC117-LS, 10-1074-LS and N-803.
Viral rebound before or at week 24 post withdrawing ART | 24 weeks
  The number of participants experiencing viral rebound, defined as confirmed HIV-1 RNA >200 copies/mL at or prior to week 24 of ART discontinuation.
ART not restarted by weeks 60 and 72 | 72 weeks
  The proportion of participants who do not meet ART restart criteria by weeks 60 and 72.
ART not restarted when bNABs below threshold | 72 weeks
  The proportion of participants who do not meet ART restart criteria for 12 or more weeks after bNAbs are below a threshold of 10 mcg/ml.

SECONDARY OUTCOMES:
Treatment-related Grade 2 adverse events | 72 weeks
  The number of participants with treatment-related solicited and unsolicited grade 2 adverse events.
Viral rebound through Step 2 | 72 weeks
  The number of participants experiencing viral rebound, defined as confirmed HIV-1 RNA >200 copies/mL, through Step 2 of the study.
Time from ART withdrawal to re-initiating ART | 72 weeks
  Time from ART withdrawal to virologic or immunologic criteria (i.e. viral load, CD4 cell count, or development of severe acute retroviral syndrome) to reinitiate ART.
Viral rebound determined by Monogram assay | 72 weeks
  Time to viral rebound (confirmed HIV-1 RNA >200 copies/mL) across different 3BNC117-LS and 10-1074-LS IC90s cut points determined by the Monogram PhenoSense assay.
Size of latent HIV-1 reservoir | 72 weeks
  Size of the latent HIV-1 reservoir, measured by IPDA and/or other appropriate assay, before, during (Step 1) and after dosing with 3BNC117-LS, 10-1074-LS and N-803 (Step 2), and after antibody concentrations have declined below a therapeutic threshold.
Changes in HIV-1 specific T Cell immune responses | 72 weeks
  Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by ELISPOT, before, during (Step 1) and after dosing with 3BNC117-LS, 10-1074-LS and N-803 (Step 2), and after antibody concentrations have declined below a therapeutic threshold.
Half-life of 3BNC117-LS and 10-1074-LS | 72 weeks
  Half-life of 3BNC117-LS and 10-1074-LS, when administered in combination with N-803 to individuals with HIV during ART interruption.
Anti-drug antibodies (ADA) | 72 weeks
  The proportion of individuals with treatment-induced ADA against each bNAb or N-803 and magnitude of the response.

OTHER OUTCOMES:
Plasma rebound virus sensitivity | 48 weeks
  The relationship between plasma rebound virus sensitivity to 3BNC117-LS and 10-1074-LS and serum levels of 3BNC117-LS and 10-1074-LS at the time of viral rebound.
HIV-1 specific T cell immune response changes | 72 weeks
  Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by assays such as polyfunctional intracellular cytokine staining (ICS) and viral inhibition assay before, during and after immunotherapy with 3BNC117-LS and 10-1074-LS in combination with N-803.
Latent HIV-1 reservoir composition | 72 weeks
  Composition of the latent HIV-1 reservoir before and after immunotherapy with 3BNC117-LS and 10-1074-LS in combination with N-803 evaluated by Q4PCR or other appropriate assays that may become available.
Neutralization sensitivity | 72 weeks
  Neutralization sensitivity by TZM/bl assay (IC50, IC80 and IC90) of representative viruses during ART and antibody suppression, and of plasma rebound viruses to 3BNC117 and 10-1074.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Caskey, MD, Principal Investigator — The Rockefeller University
Locations (3):
- United States (3):
  - Weill Cornell Medicine, Cornell Clinical Trials Unit, New York, New York
  - The Rockefeller University, New York, New York
  - Perelman School of Medicine University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No